CLINICAL TRIAL: NCT01455532
Title: A Phase 1/1b Dose Escalation Study Evaluating Iniparib (BSI201/SAR240550) as a Single Agent and in Combination With Chemotherapeutic Regimens in Patients With Solid Tumors
Brief Title: A Dose Escalation Study of Iniparib as a Single Agent and in Combination in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11746; U1111-1118-6091 (Other: UTN)
Record Dates: First submitted 2011-10-07; First posted 2011-10-20 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — iniparib; Gemcitabine; Carboplatin; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iniparib, single agent (Experimental): Iniparib will be initially administered intravenously once weekly (days 1, 8, and 15) for 3 weeks, in a 21-day cycle. Then, iniparib will be administered twice weekly (days 1, 4, 8, 11, 15, and 18) in a 21-day cycle. Cycle1 (day 1 thru day 21) will be defined as the dose limiting toxicities (DLT) observation period. Starting dose is 15 mg/kg once weekly.
  Interventions: Drug: Iniparib (SAR240550-BSI-201)
- Iniparib/Gemcitibine/Carboplatin (Experimental): Gemcitabine/carboplatin (GC) : Gemcitabine will be administered at 1,000 mg/m² as a 30min IV infusion and carboplatin area under the curve (AUC) 2 as a 60min IV infusion. Patients will receive gemcitabine/carboplatin infusions once weekly (days 1 and 8). Iniparib will be administered for two weeks, followed by a 1week of rest in a 21-day cycle (weekly schedule: days 1 and 8; twice weekly schedule: days: 1, 4, 8 and 11).
  Interventions: Drug: Iniparib (SAR240550-BSI-201); Drug: Gemcitabine; Drug: Carboplatin
- Iniparib/Paclitaxel (Experimental): Paclitaxel (P): Paclitaxel will be administered at the dose of 80 mg/m2 as a 60-minute intravenous infusion administered on days 1, 8, and 15 followed by a 1week of rest. Iniparib will be administered for three weeks, followed by 1week of rest in a 28-day cycle (weekly schedule: days 1, 8 and 15; twice weekly schedule: days 1, 4, 8, 11, 15 and 18).
  Interventions: Drug: Iniparib (SAR240550-BSI-201); Drug: Placlitaxel
- Iniparib/Pegylated liposomal doxorubicin/Carboplatin (Experimental): Pegylated liposomal doxorubicin (Doxil)/Carboplatin (PLD) : Doxil will be administered at 30 mg/m² as a 30min IV infusion and carboplatin AUC 4 as a 60min IV infusion on day 1 every four weeks. Iniparib will be administered for two weeks in a 28-day cycle (weekly schedule: days 1, and 8; twice weekly schedule: days 1, 4, 8, and 11).
  Interventions: Drug: Iniparib (SAR240550-BSI-201); Drug: Carboplatin; Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Iniparib (SAR240550-BSI-201) — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
Drug: Gemcitabine — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
  Arms: Iniparib/Gemcitibine/Carboplatin
Drug: Carboplatin — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
  Arms: Iniparib/Gemcitibine/Carboplatin; Iniparib/Pegylated liposomal doxorubicin/Carboplatin
Drug: Placlitaxel — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
  Arms: Iniparib/Paclitaxel
Drug: Pegylated liposomal doxorubicin — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
  Arms: Iniparib/Pegylated liposomal doxorubicin/Carboplatin

SUMMARY:
Primary Objective:

* To assess the safety and the maximum tolerated dose(MTD) of iniparib as a single agent and in combination with chemotherapeutic regimens in patients with advanced solid tumors that are refractory to standard therapy.

Secondary Objectives:

* To assess the antitumor effect of iniparib (per Response Evaluation Criteria in Solid Tumors [RECIST]) Version 1.1 in patients with measurable disease.
* To characterize iniparib (and its metabolites, if possible) pharmacokinetics.

Based on data generated by Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a period to assess eligibility (screening period) of up to 4 weeks (28 days), a treatment period of at least 1 cycle (3 weeks or 4 weeks depending on regimen) of study treatment, and an end-of-treatment visit at least 30 days following the last administration of study drug. However, treatment may continue until precluded by toxicity, progression, or death.

ELIGIBILITY:
Inclusion criteria:

* Capable of understanding and complying with the protocol requirements, and have signed the informed consent document
* ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* To have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic disease; that is refractory to standard therapy and/or therapies known to provide clinical benefit or for which no standard therapy exists
* For phase 1b, patients for whom the backbone chemotherapy (dose and schedule) can be considered as a standard therapeutic regime for their cancer.
* Have measurable disease or non-measurable disease, defined according to RECIST Version 1.1. Patients with skin only metastases are eligible, if the appropriate photography documentation (including measurement) of the skin metastases is provided.
* Adequate organ and bone marrow function
* Willingness, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ an effective barrier method of contraception during the study drug administration and for a period of 6 months following the last dose.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment, and at least 6 months after the last dose of study treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately. Sexually active men must agree to use a medically acceptable form of birth control during treatment and at least 6 months after the last dose. If a female partner becomes pregnant during course of study the treating physician should be informed immediately.

Exclusion criteria:

* Systemic anticancer therapy within 14 days before the first dose of study drug.
* Known allergy or hypersensitivity to components of the iniparib, gemcitabine, paclitaxel, PLD,or carboplatin formulation.
* Not recovered to Grade ≤1 from adverse events (AE), per NCI-CTCAE Version 4.03 or to within 10% of pre-treatment baseline values, due to investigational drugs, radiation, or other medications administered more than 30 days before enrollment in this study. Alopecia at screening is not exclusionary.
* Prior radical (curative) radiation therapy for treatment of cancer ≥25% of the bone marrow (1). Prior radiation to the whole pelvis is not allowed. Prior radical radiotherapy must be completed at least 4 weeks before study entry.
* Patients who have received palliative radiation therapy for symptomatic metastases must have completed treatment ≥14 days prior to initiation of study treatment.
* Active brain metastases. Patients with treated brain metastases are eligible, if 1. Radiation therapy was completed at least 2 weeks prior to study treatment; 2. Follow-up scan shows no disease progression; and 3. Patient does not require steroids. Screening for brain metastases is not required if the patient is asymptomatic.
* Clinically significant cardiac disease including congestive heart failure (New York Heart Association Class III or IV), including pre-existing ventricular arrhythmia or conduction abnormality requiring medication, or cardiomyopathy or history of a myocardial infarction within the last 6 months
* Other major medical condition (eg, uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection) which the Investigator feels might compromise the patient's effective and safe participation in the trial.
* Pregnant or breastfeeding
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or Hepatitis C Antibodies (HCAb). Testing is not required unless circumstances warrant confirmation.
* Patients with acute or chronic leukemia or with any other disease likely to have a significant bone marrow infiltration (screening not required).
* Prior treatment with gemcitabine, carboplatin, paclitaxel, or Pegylated liposomal doxorubicin.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Assessment of iniparib as single agent and in combination with chemotherapeutic agents related dose limiting toxicities (DLTs) observed at first cycle | 3 - 4 weeks

SECONDARY OUTCOMES:
To assess the antitumor effect of iniparib according to the Response Evaluation Criteria in Solid Tumors [RECIST]) Version 1.1 in patients with measurable disease | Up to 2 years
Pharmakokinetic (PK) parameters: Cmax | 0, 0.5, 1, 1.33, 1.67, 2, 4, 5, 7 and 10 h post dose
Pharmakokinetic (PK) parameters : tmax | 0, 0.5, 1, 1.33, 1.67, 2, 4, 5, 7 and 10 h post dose
Pharmakokinetic (PK) parameters: tlast | 0, 0.5, 1, 1.33, 1.67, 2, 4, 5, 7 and 10 h post dose
Pharmakokinetic (PK) parameters: AUC | 0, 0.5, 1, 1.33, 1.67, 2, 4, 5, 7 and 10 h post dose
Pharmakokinetic (PK) parameters : t1/2z | 0, 0.5, 1, 1.33, 1.67, 2, 4, 5, 7 and 10 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (6):
  - Investigational Site Number 840002, Scottsdale, Arizona
  - Investigational Site Number 840004, Los Angeles, California
  - Investigational Site Number 840010, Augusta, Georgia
  - Investigational Site Number 840007, St Louis, Missouri
  - Investigational Site Number 840001, Cincinnati, Ohio
  - Investigational Site Number 840006, San Antonio, Texas